CLINICAL TRIAL: NCT00838370
Title: Pharmacogenomic and Pharmacokinetic Safety and Cost-saving Analysis in Patients Treated With Fluoropyrimidines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Prof. dr. J.H.M. Schellens, The Netherlands Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NKI-AVL_M07PFU
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Neoplasms
Keywords: Pharmacogenetics; cost-benefit analysis; toxicity; antineoplastic drugs; Dihydropyrimidine Dehydrogenase
MeSH Terms: conditions — Neoplasms | interventions — Capecitabine; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DPYD*2A (Experimental): Patients are screened for a DPD-deficiency. Patients with a DPYD*2A mutation are eligible for intervention with capecitabine/5-FU .
  Interventions: Drug: Capecitabine, 5-fluorouracil

INTERVENTIONS:
Drug: Capecitabine, 5-fluorouracil — Patients to treat with capecitabine/5-FU will be screened prior to start of therapy for DPYD*2A. Patients heterozygous or homozygous mutant for DPYD*2A receive dose reductions of capecitabine/5-FU of at least 50% in the first two courses. In case this dose is tolerated well, doses will be increased.
  In addition, the pharmacokinetics of capecitabine/5-FU and their metabolites will be assessed in these patients.
  Other Names: Xeloda; Capecitabine; Fluorouracil; 5-Fluorouracil; 5-FU

SUMMARY:
The primary purpose of this study is to prospectively determine whether capecitabine and 5-FU-induced toxicity is preventable by dose reduction prior to start of the first administration in patients heterozygous or homozygous mutant for DPYD*2A, and to determine whether this strategy is cost-effective. Secondly, an individualized treatment algorithm for capecitabine and 5-FU therapy in DPYD*2A mutant patients will be developed and the pharmacokinetic profile of capecitabine and 5-FU will be assessed.

DETAILED DESCRIPTION:
Patients exhibiting a genetically determined disorder (DPYD*2A) in the metabolic degradation of the frequently used anticancer agents capecitabine and 5-FU (fluoropyrimidines) are at high risk of development of severe and life-threatening toxicity during standard treatment with these compounds. Treatment and recovery of this fluoropyrimidine-induced severe toxicity often requires prolonged periods of hospitalization.

Screening for DPYD*2A in patients to treat with fluoropyrimidine drugs with subsequent dose adjustments in mutant individuals prior to start of therapy will possibly reduce the number of severe toxicity events. Furthermore, by reducing the frequency and/or duration of hospitalization, substantial medical costs can be saved, making this a cost-effective strategy.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of cancer
* patient is considered for treatment with capecitabine or 5-FU
* hetero- or homozygous mutant for DPYD*2A
* able and willing to give written informed consent
* able and willing to undergo blood sampling for pharmacokinetic analysis
* life expectancy 3 months or longer
* acceptable safety laboratory values (ANC, platelet count, ASAT, ALAT, creatinine,
* WHO performance status 0-2
* no radio- or chemotherapy within the last 3 weeks prior to study entry

Exclusion Criteria:

* patients with known alcoholism, drug addiction and/or psychotic disorders that are not suitable for adequate follow-up
* women who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
safety | during fluoropyrimidine treatment of the patient

SECONDARY OUTCOMES:
cost-effectiveness | during fluoropyrimidine treatment of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Jan HM Schellens, MD, PhD, Principal Investigator — Netherlands Cancer Institute, Amsterdam, the Netherlands
Locations (3):
- Netherlands (3):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Slotervaart Hospital, Amsterdam
  - Canisius Wilhelmina Hospital, Nijmegen

REFERENCES:
- [Derived] Knikman JE, Lopez-Yurda M, Meulendijks D, Deenen MJ, Schellens JHM, Beijnen J, Cats A, Guchelaar HJ. A Nomogram to Predict Severe Toxicity in DPYD Wild-Type Patients Treated With Capecitabine-Based Anticancer Regimens. Clin Pharmacol Ther. 2024 Feb;115(2):269-277. doi: 10.1002/cpt.3100. Epub 2023 Nov 29. PMID 37957132
- [Derived] Meulendijks D, van Hasselt JGC, Huitema ADR, van Tinteren H, Deenen MJ, Beijnen JH, Cats A, Schellens JHM. Renal function, body surface area, and age are associated with risk of early-onset fluoropyrimidine-associated toxicity in patients treated with capecitabine-based anticancer regimens in daily clinical care. Eur J Cancer. 2016 Feb;54:120-130. doi: 10.1016/j.ejca.2015.10.013. Epub 2016 Jan 4. PMID 26761784
- [Derived] Deenen MJ, Meulendijks D, Cats A, Sechterberger MK, Severens JL, Boot H, Smits PH, Rosing H, Mandigers CM, Soesan M, Beijnen JH, Schellens JH. Upfront Genotyping of DPYD*2A to Individualize Fluoropyrimidine Therapy: A Safety and Cost Analysis. J Clin Oncol. 2016 Jan 20;34(3):227-34. doi: 10.1200/JCO.2015.63.1325. Epub 2015 Nov 16. PMID 26573078